CLINICAL TRIAL: NCT01166217
Title: A Phase 1, Cross-over, Single-dose, Open-label Study to Estimate the Relative Bioavailability of Three Different Formulations of Pf-04620110 Under Fed/Fasted Conditions in Healthy Adult Subjects
Brief Title: A Single Dose Study Of PF-04620110 In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B0961009
Record Dates: First submitted 2010-06-17; First posted 2010-07-20 (Estimated); Last update posted 2010-08-20 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Single Dose Study in Healthy Subjects
MeSH Terms: interventions — PF-04620110

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABCE, ACBD, BACD, BCAE, CABE and CBAD (Experimental)
  Interventions: Drug: PF-04620110

INTERVENTIONS:
Drug: PF-04620110 — The five treatments are:
  A) single dose of 5 mg immediate release tablets in the fasted state; B) single dose of 5 mg modified release osmotic capsule with a short duration of modified release 1 (MR1) in the fasted state; C) single dose of 5 mg modified release osmotic capsule with a long duration of modified release 2 (MR2) in the fasted state; D) single dose of 5 mg modified release osmotic capsule with a short duration of modified release 1 (MR1) in the fed state; E) single dose of 5 mg modified release osmotic capsule with a long duration of modified release 2 (MR2) in the fed state.

SUMMARY:
PF-04620110 is a novel compound proposed for the treatment of Type 2 diabetes mellitus. The primary purpose of this trial is to evaluate the relative bioavailability of three different oral dose formulations of PF-04620110.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 21 and 55 years
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) disease or clinical findings at screening.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Endpoints: Cmax, Tmax, AUClast, AUCinf, C24hr, peak trough ratio (PTR), and half life | following each treatment

SECONDARY OUTCOMES:
Safety Endpoints: Safety and tolerability of PF 04620110 will be assessed by physical examinations, adverse event monitoring, 12 lead electrocardiograms (ECGs), vital signs, and clinical safety laboratory measurements. | before, during and following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0961009&StudyName=A%20Single%20Dose%20Study%20Of%20PF-04620110%20In%20Healthy%20Subjects%20